CLINICAL TRIAL: NCT01094977
Title: Blood Loss and Transfusion Requirement in Infants Treated With Tranexamic Acid Undergoing Craniosynostosis Reconstruction: A Randomized Placebo-Controlled Double Blind Study of Low and High Dose Therapy
Brief Title: Blood Loss and Transfusion Requirement in Infants Treated With Tranexamic Acid
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Tara Der, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000013836
Record Dates: First submitted 2010-03-23; First posted 2010-03-29 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Craniosynostoses
Keywords: Blood Loss and Transfusion; Craniosynostoses; Tranexamic Acid; Children
MeSH Terms: conditions — Craniosynostoses; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Experimental): TXA 10mg/kg bolus before incision and 5 mg/kg infusion until skin closure
  Interventions: Drug: Tranexamic Acid
- High Dose (Experimental): TXA 100 mg/kg bolus before incision and 10 mg/kg infusion until skin closure
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Normal saline 10 ml before skin incision and infusion according to weight until skin closure
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — 10 mg/kg bolus with a 5 mg/kg/h infusion
  Arms: Low Dose
Drug: Tranexamic Acid — 100 mg/kg bolus with a 10 mg/kg/h infusion
  Arms: High Dose
Drug: Saline Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate whether tranexamic acid (TXA) reduces perioperative blood loss and transfusion requirement in infants undergoing craniosynostosis surgery.

DETAILED DESCRIPTION:
Blood loss during pediatric craniosynostosis surgery can be significant and this may be exacerbated by a dilutional coagulopathy. Multimodal blood conservation strategies may limit allogeneic transfusions, although RCTs are few and limited. It is essential to investigate these techniques to determine their potential to reduce allogeneic blood transfusions and their associated cost and morbidity.

Tranexamic acid (TXA) is a synthetic antifibrinolytic drug that competitively inhibits the lysine binding sites of plasminogen, plasmin, and tissue plasminogen activator. The result is inhibition of fibrinolysis and clot degradation.

Recent studies in adults undergoing cardiac surgery demonstrated that people with different genotypes for the plasminogen activator inhibitor-1 (PAI-1) gene may have varying degrees of bleeding. PAI-1 inhibits the transformation of plasminogen to plasmin thereby decreasing plasmin-induced fibrinolysis. Thus, PAI-1 promotes clot stability and the PAI-1 polymorphism will affect the degree of bleeding and response to TXA during craniosynostosis surgery.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 2 months to 2 years undergoing anterior cranial vault reconstruction

Exclusion Criteria:

* Known bleeding disorder as this may increase the risk of bleeding
* Current antifibrinolytic therapy as these patients may bleed less
* Patient or family history of thromboembolic disease as there may be potential risk of thrombosis
* Use of NSAIDS within 5 days of surgery as this may increase the risk of bleeding
* Known allergy to TXA
* History of renal insufficiency as TXA is renally excreted
* Acquired colour vision defects as one of the first signs of long term TXA toxicity is colour vision disturbance.

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Blood Loss | Prior and Post Surgery
  Blood loss will be carefully measured in sponges, suction cannisters, cell saver systems, and in the plastic pockets of surgical drapes.

SECONDARY OUTCOMES:
Plasminogen Activator Inhibitor-1 (PAI-1) Polymorphism - Samples | Sample will be drawn immediately after induction and prior to administration of study drug
  PAI-1 promotes clot stability and the PAI-1 polymorphism will affect the degree of bleeding and response to TXA during craniosynostosis surgery
Thromboelastography (TEG)Sample | Baseline, immediately after bolus dose of TXA is infused
  TEG monitors coagulation of blood samples in vitro to produce a complete picture of clot formation, strength and dissolution (i.e. fibrinolysis)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Der, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada